CLINICAL TRIAL: NCT03590366
Title: A Vehicle-Controlled, Double-Blind, Randomized Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects With Mild to Moderate Rosacea
Brief Title: A Study to Determine Safety and Efficacy of B244 in Subjects With Mild to Moderate Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB244-001
Record Dates: First submitted 2018-06-25; First posted 2018-07-18 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Rosacea
Keywords: Type 1 erythematotelangiectatic rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1 so that equal numbers of patients will be treated in each arm of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind study. Participants will be assigned to study treatment in accordance with the randomization schedule generated for the allocation of vehicle or B244 prior to the initiation of the trial. Randomization will be centrally-based and performed using an appropriate IWRS (an automated randomization system).
  Each participant scheduled to receive investigational product (IP) will receive a randomization number at the time of randomization. The randomization number will be used to identify the study medication kit assigned to the participant and indicate the treatment to be administered to that participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B244 (Active Comparator): B244 suspension in 30ml/bottle
  Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day.
  Interventions: Biological: B244
- Vehicle (Placebo Comparator): Vehicle, 30ml/bottle
  Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day.
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: B244 — B244 Suspension
  Arms: B244
Biological: Vehicle — Vehicle suspension
  Arms: Vehicle

SUMMARY:
This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, comparing the effect of twice daily B244 application for 8 weeks vs. vehicle application on treatment of mild to moderate rosacea.

DETAILED DESCRIPTION:
This is a Prospective, Vehicle Controlled, Double Blind, Multicenter, Randomized Phase II trial, comparing the effect of twice daily B244 application for 8 weeks vs. vehicle application on treatment of mild to moderate rosacea.

At Screening and Baseline all subjects must have Type 1 erythematotelangiectatic rosacea (ETR).

The total duration of the study will be approximately 12 weeks. Participants will report for a Screening visit and if all inclusion criteria are met will undergo a washout period, between 2 days and 4 weeks, depending on current treatment. Subjects will then report for the Baseline visit.

Subjects will come in for visits at Day 7 (Week 1), Day 28 (Week 4), and Day 56 (Week 8). A final visit will be conducted at Day 84 (Week 12).

Efficacy will be assessed using Clinician Erythema Assessment (CEA), Investigator Global Assessment (IGA), Skindex16, and Patient Self-Assessment (PSA).

Blood and urine samples will be collected for standard safety laboratory tests. Participant's safety will be monitored throughout the study.

Investigators plan to enroll approximately 130 subjects.

Randomization will be 1:1 so that equal numbers of subjects will be treated in each arm of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18.
2. A clinical diagnosis of mild to moderate facial rosacea.
3. In good general health as determined by a thorough medical history, physical examination, clinical chemistry and hematology.
4. Presence of 3 to 20 inflammatory lesions on the face (i.e. papules/pustules).
5. A Clinician Erythema Assessment (CEA) score of 2-3 at Screening and at Baseline Visits (prior to the investigational product application).
6. Mild to Moderate IGA score of 2-3 at Screening and at Baseline Visits (prior to the investigational product application).
7. Willing to refrain from using any topical or systemic treatments for the treatment of rosacea, other than the investigational product.
8. Females of childbearing potential with a negative urine pregnancy test (UPT) at Screening and Baseline/Day 1 (prior to the investigational product application).
9. Ability to comprehend and comply with study procedures.
10. Agree to commit to participate in the current protocol.
11. Provide written informed consent prior to any study procedure being performed.

Exclusion Criteria:

1. Female subjects who are pregnant, lactating or who are trying to conceive will be excluded from participation in this study.
2. Any uncontrolled chronic or serious disease or medical condition that would normally prevent participation in a clinical trial, or, in the judgment of the Investigator, would put the subject at undue risk, or might confound the study assessments (e.g., other dermatological diseases), or might interfere with the subject's participation in the study, (e.g., planned hospitalization during the study).
3. Particular forms of rosacea (e.g., rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin, Ocular rosacea Phymatous rosacea, Steroid-induced rosacea, severe rosacea including pyoderma faciale) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
4. Presence of more than two (2) nodulocystic lesions on the face.
5. Presence of less than 3 and more than 20 inflammatory lesions on the face (i.e. papules/pustules).
6. Severe papulopustular rosacea requiring systemic treatment.
7. Participation at the time of eligibility assessment (Screening) in any other investigational drug or device study or may have participated within 30 days prior to Screening.
8. Commencement of new hormonal therapy or dose change to hormonal therapy within 30 days prior to baseline. Dose and frequency of use of any hormonal therapy started more than 30 days prior to baseline must remain unchanged throughout the study. Hormonal therapies include, but are not limited to, oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (e.g. vaginal ring or transdermal hormone contraception)
9. Presence of beard or excessive facial hair at Screening which would interfere with the study treatments or study assessments and refusal to remove for duration of study.
10. Carcinoid, Pheochromocytoma or other systemic causes of flushing.
11. Known sensitivity to B244 or its components.
12. Refusal to submit to blood and urine sampling for laboratory analysis.
13. Treatment with prohibited medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ng-Cashin, MD, Study Director — Chief Medical Officer; Spiros Jamas, ScD, Study Director — AOBiome Therapeutics
Locations (9):
- United States (9):
  - Tampa Bay Medical Research, Clearwater, Florida
  - Veritas Research Corp, Miami, Florida
  - South Coast Research Center, Inc., Miami, Florida
  - FXM Research Corp., Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Paddington Testing Co., Philadelphia, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - West Houston Clinical Research Service, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- B244: B244 suspension (4x10E9 cells/ml) in 30ml/bottle
  Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day.
  B244: B244 Suspension
- Vehicle: Vehicle, 30ml/bottle
  Subjects will apply a total of 4 pumps of IP per application to the face twice-a-day.
  Vehicle: Vehicle suspension
Period: Overall Study
Arm/Group | B244 | Vehicle
Started | 73 | 67
Completed | 70 | 59
Not Completed | 3 | 8
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) Population: all subjects who all subjects who met all inclusion/exclusion criteria, were randomized, dispensed treatment, and had at least one post-treatment efficacy evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | B244 | Vehicle | Total
Number analyzed (Participants) | 73 | 67 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (15.099) | 52.4 (13.022) | 51.5 (14.120)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 48 | 103
  Male | 18 | 19 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 31 | 62
  Not Hispanic or Latino | 42 | 36 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 72 | 65 | 137
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability endpoints will consist of all treatment-related adverse events reporting during the study duration.
Time Frame: Baseline to Day 84
Population: Modified Intent to Treat (mITT) Population, which included all subjects who all subjects who met all inclusion/exclusion criteria, were randomized, dispensed treatment, and had at least one post-treatment efficacy evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 73 | 67
Participants | 5 | 6

2. Secondary Outcome: Proportion of Subjects With IGA Improvement at Week 8 Relative to Baseline.
Description: IGA (Investigator's Global Assessment) was used to assess the overall diseases severity on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild disease, 3=moderate disease, and 4=severe disease). Improvement is defined as at least 1-grade change.
Time Frame: Baseline to Day 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 73 | 67
Participants | 51 | 38

3. Secondary Outcome: Proportion of Subjects With CEA Improvement at Week 8 Relative to Baseline.
Description: Clinical Erythema Assessment (CEA) was used to assess the extent of rosacea on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). Improvement is defined as at least 1-grade change.
Time Frame: Baseline to Day 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 73 | 67
Participants | 49 | 38

4. Secondary Outcome: Change in IGA From Week 8 to Baseline.
Description: IGA (Investigator's Global Assessment) was used to assess the overall diseases severity on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild disease, 3=moderate disease, and 4=severe disease). A higher grade change indicates greater improvement in disease.
Time Frame: Baseline to Day 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 73 | 67
Participants
  Week 8 1-Grade Change | 34 | 26
  Week 8 2-Grade Change | 14 | 10
  Week 8 3-Grade Change | 3 | 2

5. Secondary Outcome: Change in CEA From Week 8 to Baseline.
Description: Clinical Erythema Assessment (CEA) was used to assess the extent of rosacea on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). A higher grade change indicates greater improvement in disease.
Time Frame: Baseline to Day 56
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 73 | 67
Participants
  Week 8 1-Grade Change | 34 | 27
  Week 8 2-Grade Change | 14 | 10
  Week 8 3-Grade Change | 1 | 1

6. Secondary Outcome: Change in Skindex 16 and Skindex 16 Sub Scores at Week 1, Week 4, Week 8 and Week 12 From Baseline.
Description: The Skindex 16 questionnaire was assigned to subjects to examine the relationship between the subject's skin health and quality of life. Subjects scored 16 questions from 0 to 6 (0=never bothered, 6=always bothered). Total scores could range between 0 to 96, where a higher score is associated with a worse quality of life.
Time Frame: Baseline to Day 84
Population: Subjects from modified Intent to Treat (mITT) Population (all subjects who all subjects who met all inclusion/exclusion criteria, were randomized, dispensed treatment, and had at least one post-treatment efficacy evaluation) that remained in the study at each respective time point for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 73 | 67
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 73 | 66
  Change from Baseline at Week 1 | -8.7 (12.584) | -12.4 (17.111)
  Change from Baseline at Week 4: number analyzed (Participants) | 71 | 59
  Change from Baseline at Week 4 | -14.5 (13.908) | -18.4 (17.418)
  Change from Baseline at Week 8: number analyzed (Participants) | 71 | 59
  Change from Baseline at Week 8 | -21.0 (20.878) | -19.9 (20.164)
  Change from Baseline at Week 12 (EOS): number analyzed (Participants) | 70 | 59
  Change from Baseline at Week 12 (EOS) | -19.7 (22.152) | -20.6 (22.694)

7. Secondary Outcome: Proportion of Subjects With Change in PSA at Week 1, Week 4, Week 8 and Week 12 From Baseline.
Description: Subjects were asked to perform static ("snap-shot") evaluations of their rosacea-associated facial erythema severity using the Patient Self Assessment scale (PSA) at each study visit, and report the one integer that best describes the overall severity of their facial redness as seen in a mirror at the time of the evaluation on a scale of 0 to 4 (0=no redness, 1=very mild redness, 2=mild redness, 3=moderate redness, 4=severe redness). A higher grade change indicates greater improvement.
Time Frame: Baseline to Day 84
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | B244 | Vehicle
Number analyzed (Participants) | 73 | 67
Participants
  Week 1: number analyzed (Participants) | 73 | 66
  Week 1: 0-Grade Change | 49 | 44
  Week 1: 1-Grade Change | 19 | 19
  Week 1: 2-Grade Change | 5 | 3
  Week 1: 3-Grade Change | 0 | 0
  Week 4: number analyzed (Participants) | 71 | 59
  Week 4: 0-Grade Change | 29 | 23
  Week 4: 1-Grade Change | 36 | 30
  Week 4: 2-Grade Change | 5 | 6
  Week 4: 3-Grade Change | 1 | 0
  Week 8: number analyzed (Participants) | 71 | 59
  Week 8: 0-Grade Change | 23 | 21
  Week 8: 1-Grade Change | 31 | 24
  Week 8: 2-Grade Change | 14 | 11
  Week 8: 3-Grade Change | 3 | 3
  Week 12 (EOS): number analyzed (Participants) | 70 | 59
  Week 12 (EOS): 0-Grade Change | 23 | 22
  Week 12 (EOS): 1-Grade Change | 29 | 21
  Week 12 (EOS): 2-Grade Change | 15 | 14
  Week 12 (EOS): 3-Grade Change | 3 | 2

ADVERSE EVENTS:
Time Frame: Baseline to Week 12.
Description: Beginning with the Screening visit and through the end of study or early termination (ET) visit, the PI and study personnel reviewed each subject's clinical evaluation findings and queried the subject directly regarding AEs. Subjects were to be followed for AEs until 30 days post study conclusion or until the PI determined the AEs were stable, whichever was later. PIs monitored each subject for clinical evidence of adverse events on a routine basis throughout the study.
Arm/Group | B244 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/67
Other Adverse Events (participants affected / at risk) | 19/73 | 12/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 (N=73) | Vehicle (N=67)
Hordeolum (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Application site pain (General disorders) | 1 | 3
Application site dryness (General disorders) | 1 | 2
Application site pruritus (General disorders) | 0 | 2
Application site erythema (General disorders) | 0 | 1
Application site plaque (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dermatitis contact (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have 60 days to review the papers. Sponsor shall have the right to require Institution/Principal Investigator, as applicable, to remove specifically identified confidential information and/or delay the proposed publication or presentation for an additional 90 days to enable Sponsor to seek patent protections.

DOCUMENTS (2):
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT03590366/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT03590366/SAP_001.pdf